CLINICAL TRIAL: NCT04608435
Title: Sex Differences in Postoperative Sleep Quality and Inflammation in Patients Undergoing Video-Assisted Thoracoscopic Surgery
Brief Title: Sex Differences in Postoperative Sleep Quality and Inflammation
Status: Completed | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, principal investigator, Shengjing Hospital
Other Study IDs: Sex, sleep and inflammation
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Sex Differences; Postoperative Sleep Quality; Postoperative Pain; Inflammation Function
Keywords: sex differences; postoperative sleep quality; postoperative pain; inflammation function
MeSH Terms: conditions — Pain, Postoperative | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male Group
  Interventions: Other: Video-Assisted Thoracoscopic Surgery
- Female Group
  Interventions: Other: Video-Assisted Thoracoscopic Surgery

INTERVENTIONS:
Other: Video-Assisted Thoracoscopic Surgery — patients receive Video-Assisted Thoracoscopic Surgery under general anesthesia

SUMMARY:
Video-Assisted Thoracoscopic Surgery(VATS) is among the most common and disabling persistent pain and inflammation conditions, with increasing prevalence in the developed world, and affects women to a greater degree than men. And sleep disruption also remains a challenging problem in surgical settings. Postoperative sleep disturbances (POSD) are defined as changes in the sleep structure and quality of patients during the early stages after surgery, which are manifested as significantly shortened rapid eye movement (REM) sleep, prolonged awake time, and sleep fragmentation. Long-term POSD may increase the risk of postoperative delirium or cognitive dysfunction and delay recovery, thereby worsening the patient's physical condition. The aim of the study was to investigate the effect of sex differences on postoperative pain, inflammation and sleep quality among patients who have undergone video-assisted thoracoscopic surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* ASA I-III
* under general anesthesia

Exclusion Criteria:

* patients with central nervous system and mental diseases;
* patients with preoperative sleep disturbances;
* patients with a history of sedative, analgesic, or antidepression drug use;
* patients with sleep apnea or moderate and severe obstructive sleep apnea-hypopnea syndrome;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing video-assisted thoracoscopic surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2020-10-31 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
sleep quality of one night before surgery | first night before surgery
  Use Athens insomnia scale to test the sleep quality the first night before surgery
sleep quality of first night after surgery | first night after surgery
  Use Athens insomnia scale to test the sleep quality the first night after surgery
sleep quality of third night after surgery | third night after surgery
  Use Athens insomnia scale to test the sleep quality the third night after surgery

SECONDARY OUTCOMES:
visual analog scale(VAS) score after surgery | one day before surgery
  evaluate VAS score after surgery
visual analog scale(VAS) score after surgery | 3 hours after surgery
  evaluate VAS score after surgery
visual analog scale(VAS) score after surgery | 8 pm the first day after surgery
  evaluate VAS score after surgery
postoperative adverse effect | 24 hours after surgery
  evaluate postoperative adverse effect 24 hours after surgery
perioperative inflammation function | two days before surgery
  evaluate neutrophils
perioperative inflammation function | two days before surgery
  evaluate platelet
perioperative inflammation function | two days before surgery
  evaluate lymphocyte
perioperative inflammation function | first days after surgery
  evaluate neutrophils,platelet,lymphocyte
perioperative inflammation function | first days after surgery
  evaluate neutrophils
perioperative inflammation function | first days after surgery
  evaluate platelet
perioperative inflammation function | first days after surgery
  evaluate lymphocyte
Postoperative cognition evaluation | one day before surgery
  Use MMSE Mini-Mental State Examination (MMSE) was also evaluated at Sleep preop 1, Sleep POD 1 and Sleep POD 3.18 Each correct answer is 1 point, and error or unknown is 0 point. The unsuitable one is 9 points, and refusing to answer or incomprehension is 8 points. In the total score, 8 points and 9 points are calculated by 0 points. The highest score is 30 points. The division of dementia or not is related to the degree of education. The dementia is affirmed by the patient who is illiterate and less than 17 points, the primary school is less than 20 points, and more than middle school is less than 24 points. The scores which from 27 to 30 is normal, 21 to 26 of mild, 10 to 20 of moderate, and from 0 to 9 is severe.
Postoperative cognition evaluation | first day after surgery
  Use MMSE Mini-Mental State Examination (MMSE) was also evaluated at Sleep preop 1, Sleep POD 1 and Sleep POD 3.18 Each correct answer is 1 point, and error or unknown is 0 point. The unsuitable one is 9 points, and refusing to answer or incomprehension is 8 points. In the total score, 8 points and 9 points are calculated by 0 points. The highest score is 30 points. The division of dementia or not is related to the degree of education. The dementia is affirmed by the patient who is illiterate and less than 17 points, the primary school is less than 20 points, and more than middle school is less than 24 points. The scores which from 27 to 30 is normal, 21 to 26 of mild, 10 to 20 of moderate, and from 0 to 9 is severe.
Postoperative cognition evaluation | third day after surgery
  Use MMSE Mini-Mental State Examination (MMSE) was also evaluated at Sleep preop 1, Sleep POD 1 and Sleep POD 3.18 Each correct answer is 1 point, and error or unknown is 0 point. The unsuitable one is 9 points, and refusing to answer or incomprehension is 8 points. In the total score, 8 points and 9 points are calculated by 0 points. The highest score is 30 points. The division of dementia or not is related to the degree of education. The dementia is affirmed by the patient who is illiterate and less than 17 points, the primary school is less than 20 points, and more than middle school is less than 24 points. The scores which from 27 to 30 is normal, 21 to 26 of mild, 10 to 20 of moderate, and from 0 to 9 is severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No